CLINICAL TRIAL: NCT04174586
Title: Cord Blood Microtransplantation for Treatment of Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-001
Record Dates: First submitted 2019-10-14; First posted 2019-11-22 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Safety Issues; Efficiency
Keywords: Cord blood microtransplatation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cord blood group (Experimental): standard induction and consolidation chemotherapy with cord blood microtransplantation
  Interventions: Biological: microtransplantation

INTERVENTIONS:
Biological: microtransplantation — HLA mismatched donor cord blood infusion

SUMMARY:
Discuss the effectiveness and safety of cord blood microtransplantation for treatment of acute myeloid leukemia

DETAILED DESCRIPTION:
The investigators conducted a prospective, single center clinical trial to dissuss the outcomes and toxicities of HLA-mismatched cord blood infusion after chemotherapy (microtransplantation) in older patients with acute myeloid leukemia (AML)

ELIGIBILITY:
Inclusion Criteria:

1. de novo acute myeloid leukemia
2. age 60-80

Exclusion Criteria:

1. have no suitable donor or donor refused
2. patient refused to accept donor cells

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 1 month
  Bone marrow <5% blasts； Absolute neutrophil count >1000/mcL； Platelets ≥100,000/mcL；No residual evidence of extramedullary disease.
time of hematopoietic recovery | 1 month
  Absolute neutrophil count >500/mcL; Platelets ≥20,000/mcL

SECONDARY OUTCOMES:
time to progression | 2 year
  Measured from complete remission to the relapse

OTHER OUTCOMES:
diease free survival | 2 year
  Measured from complete remission to the date of death or the date of last follow-up examination.
overall survival | 2 year
  Measured from the date of beginning therapy to the date of death or the date of last follow-up examination.
rate of early mortality | 1 month
  Death within 4 weeks after initiation of induction therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zimin Sun, Study Chair — The First Affiliated Hospital of USTC
Locations (1):
- The First Affiliated Hospital of USTC, Hefei, China